CLINICAL TRIAL: NCT01547780
Title: PET Imaging of Translocator Protein in Subjects With Traumatic Brain Injury
Brief Title: Translocator Protein and Inflammation After Traumatic Brain Injury
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Collaborators: Suburban Hospital (Other); Uniformed Services University of the Health Sciences (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 120063; 12-M-0063
Record Dates: First submitted 2012-03-06; First posted 2012-03-08 (Estimated); Results first posted 2021-07-30 (Actual); Last update posted 2021-07-30 (Actual); Status verified 2017-09-28

CONDITIONS: Traumatic Brain Injury (TBI); Healthy
Keywords: Positron Emission Tomography (PET); Inflammation; Microglial Activation; Traumatic Brain Injury; TBI
MeSH Terms: conditions — Brain Injuries, Traumatic; Inflammation | interventions — (methyl-(11)C)N-acetyl-N-(2-methoxybenzyl)-2-phenoxy-5-pyridinamine; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Baseline brain PET in acute TBI patient (Experimental): Single intravenous injection of [C-11]PBR28, ~10-20 mCi, prior to baseline brain positron emission tomography (PET) scan in Acute (< 5 months post-injury) traumatic brain injury (TBI) patients.
  Interventions: Drug: [11C]PBR28 and Positron Emission Tomography (PET)
- Repeat brain PET in acute TBI patient (Experimental): Single intravenous injection of [C-11]PBR28, ~10-20 mCi, prior to repeat brain positron emission tomography (PET) scan in Acute (< 5 months post-injury) traumatic brain injury (TBI) patients.
  Interventions: Drug: [11C]PBR28 and Positron Emission Tomography (PET)
- Single brain PET in Chronic TBI patient (Experimental): Single intravenous injection of [C-11]PBR28, ~10-20 mCi, prior to brain positron emission tomography (PET) scan in Chronic (5 months - 5 years post-injury) traumatic brain injury (TBI) patients.
  Interventions: Drug: [11C]PBR28 and Positron Emission Tomography (PET)
- Single brain PET in healthy subjects (Experimental): Single intravenous injection of [C-11]PBR28, ~10-20 mCi, prior to brain positron emission tomography (PET) scan in Healthy Subjects.
  Interventions: Drug: [11C]PBR28 and Positron Emission Tomography (PET)

INTERVENTIONS:
Drug: [11C]PBR28 and Positron Emission Tomography (PET) — Brain PET with [11C]PBR28. 11C]PBR28 is a new PET ligand that images TSPO with high levels of specific binding.

SUMMARY:
Background:

- People with traumatic brain injury (TBI) often have inflammation in the brain. A protein called the translocator protein (TSPO) is often present with inflammation. Researchers want to see if a radioactive chemical known as [11C]PBR28 can be used to study TSPO and inflammation in the brain of people with TBI.

Objectives:

- To test whether [11C]PBR28 can be used to study changes in the brain after a traumatic brain injury.

Eligibility:

* Individuals at least 18 years of age who have had TBI and have had a brain scan that shows signs of inflammation.
* Healthy volunteers at least 18 years of age.

Design:

* Participants will be screened with a physical exam and medical history. Blood and urine samples will be collected.
* All participants will have two brain scans during an outpatient visit. A magnetic resonance imaging scan will study brain activity. A positron emission tomography (PET) scan will use [11C]PBR28 to look for signs of TSPO and brain inflammation.
* Participants with TBI will have two PET scans within 10 days of the head injury, and a PET scan around 90 days after the injury. They may also have MRI scans under this or another study. Tests of thinking, memory, and concentration will be used to study the effects of the injury and inflammation

DETAILED DESCRIPTION:
Objective:

Brain damage following traumatic injury (TBI) results from both direct (e.g., mechanical injury to the brain and vasculature) and indirect mechanisms (e.g., secondary mechanisms such as inflammation). While CT and MRI can help visualize the result of inflammatory processes in the brain for instance, the development of cerebral edema neither method can be used to document active inflammation itself. The translocator protein (TSPO), which is highly expressed in microglia and reactive astrocytes, has been used as a biomarker in positron emission tomography (PET) to identify active inflammatory processes. Recently, our laboratory developed PBR28, a new PET ligand that images TSPO with high levels of specific binding. We have successfully used PBR28 to investigate a number of brain disorders such as epilepsy, multiple sclerosis, and HIV infection with minor cognitive motor disorder, and are detecting neuroinflammation. The current protocol aims to explore whether PBR28 PET imaging can show changes in subjects with TBI who have shown MRI abnormalities in the acute phase and also in those who are in the chronic phase of TBI.

Study population: The following three groups will be studied:

TBI subjects who had brain injury within approximately 3 months and have exhibited MRI abnormalities consistent with TBI and who are enrolled in "Evaluation, Pathogenesis, and Outcome of Subjects with or Suspected Traumatic Brain Injury" (10-N-N122, PI Latour), "Evaluation and Diagnosis of Potential Research Subjects with Traumatic Brain Injury (TBI), (11-N-0084, PI: Lawrence Latour), or other CNRM protocols. N = 20

TBI subjects who had brain injury more than approximately 5 month ago, are enrolled in 11-N-0084, and meet criteria of TBI established by CNRM. N = 20

Healthy age-matched volunteers. N = 20.

Design:

This is an exploratory study to determine whether PBR28 can detect the increased TSPO associated with neuroinflammation by scanning subjects who have shown MRI abnormalities in the acute phase. We also investigate whether PBR28 detects changes in the chronic phase as recently reported using an old ligand, PK 11195. Two groups of TBI subjects will be studied depending on their availability relative to the time of injury. To investigate changes in TSPO in the areas of MRI abnormalities in the acute phase, one group of TBI subjects (n = 20) will be studied who have shown TBI- related MRI abnormalities. These participants will have up to four PBR28 PET scans; one to two PET scans within approximately 10 days of head injury, a third PET scan approximately three months after injury, and a fourth scan approximately one year after the scan at ~three months. To study changes in TSPO in the chronic phase, another group of TBI subjects will be enrolled who had brain injury more than approximately 5 months but within 5 years ago and meet the criteria of TBI by CNRM. This separate group is included because some TBI subjects are being recruited by CNRM only sometime after the injury. The participants at the chronic phase will have one PET and one MRI scan. In addition to MRI data, for all TBI subjects, clinical information obtained in 10-N-N122 (only the acute phase) and 11-N-0084 (both acute and chronic phase) will be used to evaluate the utility of the PET data in order to better understand the pathology of TBI.

Outcome Measures:

In this exploratory study to investigate the ability of PBR28 PET to detect increases in TSPO, the primary goal will be to measure the magnitude and variance of any increases observed in PBR28 binding in areas of inflammation following TBI. Those data may be used to design future studies with a larger sample size.

ELIGIBILITY:
-INCLUSION CRITERIA:

Subjects with TBI:

Subjects with TBI eligible for participation in this research study must meet the following inclusion criteria. Depending on the timing of the availability of the subjects the following two groups will be studied. No subject will be enrolled in both group 1 and 2.

Group 1 Acute/subacute phase (n = 20)

* Diagnosis of non-penetrating TBI caused by a head injury within approximately 5 months.
* Ambulatory.
* Able to provide self consent without a legally-authorized representative based on the assessment of the Decision-Making Capacity (DMC) by the Human Subjects Protection Unit (HSPU).
* Show abnormal MRI findings consistent with TBI in protocol 10-N-N122 or in the image database of the CNRM Image Processing Core if the subject is recruited from CNRM Recruitment Core protocol 11-N-0084 or another CNRM protocol that allows referrals to other studies.
* Age 18 or older.

Group 2 Chronic phase (n = 20)

* A head injury approximately 5 months 5 years ago.
* Enrolled in CNRM Recruitment Core protocol 11-N-0084 or another CNRM protocol that allows referral to other studies.
* Meet at least one of the criteria of Probable or Definite TBI established by CNRM.
* Ambulatory.
* Able to provide self consent without a legally-authorized representative based on the assessment of the Decision-Making Capacity (DMC) by the Human Subjects Protection Unit (HSPU).
* Age 18 or older.

Group 3 Healthy subjects.

* Healthy without past or present history of brain disease.
* Age 18 or older.

EXCLUSION CRITERIA:

Subjects with TBI for both groups 1 and 2 are not eligible for participation in this research study if any of the following conditions exist:

1. Present or past history of brain disease other than TBI.
2. Subjects with abnormal MRI findings that suggest a diagnosis other than TBI or a second lesion such as brain tumor in addition to the changes consistent with TBI.
3. Serious medical conditions, which make study procedures of the current study unsafe. Such serious medical conditions include uncontrolled epilepsy and multiple serious injuries. The Medical Advisory Investigator of this protocol will determine whether the subject needs to be excluded.
4. Contraindication to MRI scanning including certain metal implants or devices such as: cardiac pacemaker, insulin infusion pump, implanted drug infusion device, cochlear, otologic, or ear implant, transdermal medication patch (Nitroglycerine) that cannot be removed for the study, body piercing(s), bone/joint pin, screw, nail, plate, wire sutures or surgical staples, shunts, cerebral aneurysms clips, shrapnel or other metal imbedded in a subject's body (such as from war wounds or accidents or previous work in metal fields or machines that may have left any metallic fragments in or near the subject's eyes).
5. Conditions precluding entry into the scanners (e.g. morbid obesity, claustrophobia, etc.).
6. In female subjects, pregnancy or breastfeeding.
7. Exposure to research related radiation in the past year that, when combined with this study, would place subjects above the allowable limits.

HEALTHY SUBJECTS ARE NOT ELIGIBLE FOR PARTICIPATION IN THIS RESEARCH IF ANY OF THE FOLLOWING CONDITIONS EXIST:

1. Any past or present history of DSM Axis I disorder, with the exception of substance abuse that ended over 6 months prior to enrollment.
2. Contraindication to MRI scanning including certain metal implants or devices such as: cardiac pacemaker, insulin infusion pump, implanted drug infusion device, cochlear, otologic, or ear implant, transdermal medication patch (Nitroglycerine) that cannot be removed for the study, body piercing(s), bone/joint pin, screw, nail, plate, wire sutures or surgical staples, shunts, cerebral aneurysms clips, shrapnel or other metal imbedded in a subject's body (such as from war wounds or accidents or previous work in metal fields or machines that may have left any metallic fragments in or near the subject's eyes).
3. Conditions precluding entry into the scanners (e.g. morbid obesity, claustrophobia, etc.).
4. In female subjects, pregnancy or breastfeeding.
5. Clinically significant laboratory abnormalities, as defined as laboratory values that are out of normal range or require clinical workup and/or treatment.
6. Exposure to research related radiation in the past year that, when combined with this study, would place subjects above the allowable limits.
7. Previously determined as a low-affinity binder in another study on TSPO.
8. Positive results of urine drug screen on enrollment.

HIV positive subjects are considered healthy as long as he/she does not show neurological or psychiatric symptoms based on history and physical exams. Results of HIV test in both TBI subjects and healthy controls may help interpretation of the PET results. Statistical analysis: Analysis of date/study outcomes. Results of urine drug screen and history of using drugs of abuse may also help interpretation of the PET results. In addition, inclusion of TBI subjects who show positive for urine drug screen may improve recruitment of TBI subjects.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2012-01-20; Primary Completion 2017-09-28 (Actual); Study Completion 2017-09-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Innis, MD, PhD, Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Brown AK, Fujita M, Fujimura Y, Liow JS, Stabin M, Ryu YH, Imaizumi M, Hong J, Pike VW, Innis RB. Radiation dosimetry and biodistribution in monkey and man of 11C-PBR28: a PET radioligand to image inflammation. J Nucl Med. 2007 Dec;48(12):2072-9. doi: 10.2967/jnumed.107.044842. Epub 2007 Nov 15. PMID 18006619
- [Background] Cernak I, O'Connor C, Vink R. Activation of cyclo-oxygenase-2 contributes to motor and cognitive dysfunction following diffuse traumatic brain injury in rats. Clin Exp Pharmacol Physiol. 2001 Nov;28(11):922-5. doi: 10.1046/j.1440-1681.2001.03549.x. PMID 11703397
- [Background] Conzen M, Ebel H, Swart E, Skreczek W, Dette M, Oppel F. Long-term neuropsychological outcome after severe head injury with good recovery. Brain Inj. 1992 Jan-Feb;6(1):45-52. doi: 10.3109/02699059209008121. PMID 1739852
- [Derived] Paul S, Gallagher E, Liow JS, Mabins S, Henry K, Zoghbi SS, Gunn RN, Kreisl WC, Richards EM, Zanotti-Fregonara P, Morse CL, Hong J, Kowalski A, Pike VW, Innis RB, Fujita M. Building a database for brain 18 kDa translocator protein imaged using [11C]PBR28 in healthy subjects. J Cereb Blood Flow Metab. 2019 Jun;39(6):1138-1147. doi: 10.1177/0271678X18771250. Epub 2018 May 11. PMID 29749279

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 52 subjects were consented but two subjects withdrew after consent/lost to follow up.
Groups:
- Baseline Brain PET in Acute TBI Patient: One ~10-20 mCi intravenous injection of [C-11]PBR28 prior to baseline brain positron emission tomography (PET) scan in Acute (< 5 months post-injury) traumatic brain injury (TBI) patients.
- Single Brain PET in Chronic TBI Patient: One ~10-20 mCi intravenous injection of [C-11]PBR28 prior to brain positron emission tomography (PET) scan in Chronic (5 months - 5 years post-injury) traumatic brain injury (TBI) patients.
- Single Brain PET in Healthy Subjects: One ~10-20 mCi intravenous injection of [C-11]PBR28 prior to brain positron emission tomography (PET) scan in Healthy Subjects.
Period: Baseline PET Scan
Arm/Group | Baseline Brain PET in Acute TBI Patient | Repeat Brain PET in Acute TBI Patient | Single Brain PET in Chronic TBI Patient | Single Brain PET in Healthy Subjects
Started | 12 | 0 | 19 | 19
Completed | 9 | 0 | 17 | 19
Not Completed | 3 | 0 | 2 | 0
Not completed — Physician Decision | 1 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 1 | 0
Period: Repeat PET Scan
Arm/Group | Baseline Brain PET in Acute TBI Patient | Repeat Brain PET in Acute TBI Patient | Single Brain PET in Chronic TBI Patient | Single Brain PET in Healthy Subjects
Started (Period 2 only applicable to repeat PET Scan) | 0 | 4 | 0 | 0
Completed | 0 | 4 | 0 | 0
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Baseline Brain PET in Acute TBI Patient | Single Brain PET in Chronic TBI Patient | Single Brain PET in Healthy Subjects | Total
Number analyzed (Participants) | 12 | 19 | 19 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 0 | 1
  Between 18 and 65 years | 7 | 17 | 16 | 40
  >=65 years | 4 | 2 | 3 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 6 | 7 | 14
  Male | 11 | 13 | 12 | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 2 | 6
  Not Hispanic or Latino | 10 | 17 | 17 | 44
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 5 | 4 | 4 | 13
  White | 5 | 14 | 14 | 33
  More than one race | 0 | 1 | 0 | 1
  Unknown or Not Reported | 2 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Receptor Binding (Vt)
Description: To determine total distribution volume of [C-11]PBR28 in the whole brain using PET and arterial input function (concentration of radioligand in arterial plasma over time).
Time Frame: 120 minutes from the start of the PET scan
Population: The analyses only included subjects who completed the brain [C-11]PBR28 PET scan
Measure: Mean (Standard Deviation); unit: mL/cm^3
Arm/Group | Baseline Brain PET in Acute TBI Patient | Repeat Brain PET in Acute TBI Patient | Single Brain PET in Chronic TBI Patient | Single Brain PET in Healthy Subjects
Number analyzed (Participants) | 7 | 3 | 16 | 16
mL/cm^3 | 2.53 (0.50) | 2.21 (0.49) | 3.21 (1.04) | 3.22 (0.81)

2. Primary Outcome: Receptor Binding Corrected for Plasma (Vt/fp)
Description: Total distribution volume divided by plasma free fraction (fp) of [C-11]PBR28. Measured with PET and arterial input function (concentration of radioligand in arterial plasma over time).
Time Frame: 120 minutes from the start of the PET scan
Population: The analyses only included subjects who completed the brain [C-11]PBR28 PET scan
Measure: Mean (Standard Deviation); unit: mL/cm^3
Arm/Group | Baseline Brain PET in Acute TBI Patient | Repeat Brain PET in Acute TBI Patient | Single Brain PET in Chronic TBI Patient | Single Brain PET in Healthy Subjects
Number analyzed (Participants) | 7 | 3 | 16 | 16
mL/cm^3 | 93.72 (20.83) | 80.32 (10.35) | 118.73 (37.98) | 103.99 (29.52)

ADVERSE EVENTS:
Time Frame: 24 hours
Arm/Group | Baseline Brain PET in Acute TBI Patient | Repeat Brain PET in Acute TBI Patient | Single Brain PET in Chronic TBI Patient | Single Brain PET in Healthy Subjects
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/4 | 0/19 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/4 | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 0/12 | 0/4 | 0/19 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-10): https://cdn.clinicaltrials.gov/large-docs/80/NCT01547780/Prot_SAP_000.pdf